CLINICAL TRIAL: NCT05433714
Title: The Reliability and Validity of the Figure of 8 Walk Test in Multiple Sclerosis
Brief Title: Figure of 8 Walk Test in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, Zekiye İpek KATIRCI KIRMACI, Asst. Prof., Kahramanmaras Sutcu Imam University
Other Study IDs: ipekkrmc
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Multiple Sclerosis
Keywords: multiple scleorsis; balance; Walking
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple sclerosis patient: First day, first evaluator will perform all tests, and second day, second evaluator will perform the figure of 8 walk test.
  Interventions: Other: Assesment

INTERVENTIONS:
Other: Assesment — The figure of walk test, Berg Balance scale, Timed 25-Foot Walk, Timed up and go test, Foursquare walk test

SUMMARY:
Balance disorder is common in people with MS. As the disease worsens, it is associated with impaired balance, difficulty walking, decreased mobility, and an increased risk of falling. Given the prevalence and clinical significance of balance dysfunction in individuals with MS, the assessment of balance has become an important focus in MS clinical practice and research. The figure of 8 Walk Test is a standard clinical measure used to evaluate the forward walking performance required in daily life. Beyond walking straight, turning ability is required in many situations in daily life such as walking around a table, avoiding obstacles and navigating the street. The gait characteristics of walking on a straight and curved road are different. During curved walking, the center of mass of the body shifts to the inner leg as the stance time of the inner leg increases, as opposed to walking on a straight track. Compared to other standardized tests, scoring is not dependent on the subjectivity of the examiner, can be administered by a person with minimal training, and requires minimal time, space, and equipment. The test assesses the ability to quickly change direction of movement and is a timed test involving the use of assistive devices.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a progressive disease of the central nervous system characterized by demyelination and destruction of motor and sensory axons. As the disease worsens, it is associated with impaired balance, difficulty walking, decreased mobility, and an increased risk of falling. The prevalence of balance dysfunction in individuals with MS and Given its clinical relevance, the assessment of balance has become an important focus in MS clinical practice and research. The figure of 8 Walk Test is a standard clinical measure used to evaluate the forward walking performance required in daily life.In the figure of 8 walk test, two cones are placed 1.5 meters apart. The individual stands in the middle of this distance. At the start of the test, he goes around the first cone as fast as he can walk around the first cone, then when he comes to the other starting point, this time around the other cone. The elapsed time is recorded.

The aim of the study is to examine the validity and reliability of the 8-shape walking test in MS patients.

ELIGIBILITY:
Inclusion Criteria:

* Having an EDSS score of 4 and below,
* Being between the ages of 18-65
* Willingness to participate in the study

Exclusion Criteria:

* Being pregnant or within the first 3 months after giving birth,
* Receiving corticosteroid therapy in the last 1 month,
* Using drugs that will affect walking in the last 1 month

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis Patients
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
The Figure of Walk Test | First day
  Two cones are placed 1.5 meters apart. The individual stands in the middle of this distance. At the start of the test, he goes around the first cone as fast as he can walk around the first cone, then when he comes to the other starting point, this time around the other cone. Elapsed time is recorded
The Figure of Walk Test | second day
  Two cones are placed 1.5 meters apart. The individual stands in the middle of this distance. At the start of the test, he goes around the first cone as fast as he can walk around the first cone, then when he comes to the other starting point, this time around the other cone. Elapsed time is recorded

SECONDARY OUTCOMES:
Berg Balance scale | First day
  It is a 14-item scale that measures the ability to maintain balance while performing functional tasks. Each item is scored between 0 and 4. Balance is considered good if the total score is 45 and above.
Timed up and go test | First day
  At the beginning of the test, individuals sit in a chair. A distance of 3 m is set in front of it. With the start command, he gets up from his seat and walks 3 m, turns around and walks back and sits. With the start command, the time to sit on the chair is recorded in seconds. Short duration indicates good functional mobility.
Timed 25-Foot Walk test | First day
  It is an evaluation to evaluate mobility and leg functions. Individuals are asked to safely walk 7.62 m on a flat surface at their highest speed.
Four Square Step Test | First day
  It aims to assess dynamic balance and step objects forward, sideways and backwards. The square drawn on the floor is divided into 4 equal parts. The number 1 is written in the lower right corner, up to 4 clockwise. With the start command, individuals are asked to step on the numbers in order.

CONTACTS AND LOCATIONS:
Overall Officials: Zekiye İpek Katırcı Kırmacı, Principal Investigator — Kahramanmaras Sutcu Imam University
Locations (1):
- Kahramanmaraş Sutcu Imam University, Kahramanmaraş, Turkey (Türkiye)